CLINICAL TRIAL: NCT04607811
Title: Using Behavioral Economics to Improve Mobility for Adults With Stroke
Brief Title: Behavioral Economics and Mobility After Stroke (BE Mobile)
Acronym: BE Mobile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 843894
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Stroke
Keywords: physical activity; wearable; gamification
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Participants will wear the Fitbit device and record their daily step counts during the baseline and 8 week intervention period. Participants will complete study surveys at baseline and the end of the 8 week intervention.
- Gamification arm (Experimental): Participants will wear the Fitbit device and record their daily step counts during the baseline and 8 week intervention period. Participants will have a weekly step goal they are encouraged to meet. Participants will engage in a social incentive-based gamification based on points and levels that leverages loss aversion, which has been demonstrated to motivate behavior change more effectively with losses than gains. Participants will receive daily feedback for the step counts and weekly feedback for levels. Participants will be asked to identify a support partner, who will receive weekly reports with the the participant's points and levels balance.
  Interventions: Behavioral: Gamification with social incentives

INTERVENTIONS:
Behavioral: Gamification with social incentives — Participants will select a step goal that is 33%, 40%, or 50% above their baseline step value. Participants in this group will participate in a game with points and levels to help motivate participants to meet their daily step goal. Additionally, all participants will identify a support partner to receive weekly updates on their performance and offer positive encouragement to help the participant meet their step goal.
  Arms: Gamification arm

SUMMARY:
In this pilot, randomized controlled trial, the investigators will compare the preliminary effectiveness of a gamification with social incentives 8 week intervention to increase physical activity for adults with stroke.

DETAILED DESCRIPTION:
In this 2 arm randomized trial, the investigators will compare the preliminary effectiveness of a social incentive-based gamification intervention to increase physical activity relative to a control arm among adults with stroke. All participants will use a Fitbit wearable device to establish a baseline step count, select a step goal increase of 33% to 50% above their baseline and then participate in an 8 week intervention. The gamification arm will be entered into a game with points and levels designed using insights from behavioral economics. They will be asked to select a social support partner who will receive weekly updates on their progress in the game.

ELIGIBILITY:
Inclusion Criteria:

* History of ischemic or hemorrhagic stroke (confirmed with ICD-10 or DRG code) at least 3 months prior to enrollment
* Ability to provide informed consent
* Life Space Assessment mobility level 3
* Ability to ambulate outside of their home (self-reported)
* Owns a smartphone or tablet compatible with required applications for the wearable tracking device
* Sufficient cognitive ability to participate (5-minute Montreal Cognitive Assessment Score ≥ 11 points)

Exclusion Criteria:

* Inability to provide informed consent, illiteracy or inability to speak, read, and write English
* Self-reported history of falls within the last 3 months
* Severe cognitive impairment (MoCA score ≤ 10 points)
* Medical condition that may limit participation in physical activity program (e.g. metastatic cancer, end-stage renal disease)
* Currently institutionalized in skilled nursing or long-term care facility
* Baseline step count > 7500/day
* Currently receiving physical therapy services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Daily step counts | Intervention weeks 1-8
  Change in mean daily steps from baseline

SECONDARY OUTCOMES:
Daily step counts | Intervention weeks 1-8
  Proportion of days participants in the gamification arm met their daily step goal

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Greysen, MD, MHS, MA, Principal Investigator — University of Pennsylvania; Kimberly J Waddell, PhD, MS, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waddell KJ, Patel MS, Clark K, Harrington TO, Greysen SR. Leveraging insights from behavioral economics to improve mobility for adults with stroke: Design and rationale of the BE Mobile clinical trial. Contemp Clin Trials. 2021 Aug;107:106483. doi: 10.1016/j.cct.2021.106483. Epub 2021 Jun 12. PMID 34129953